CLINICAL TRIAL: NCT05419895
Title: Early Diagnostic Response Model (EDRM): Evaluating an Early Screening to Evaluation Pilot Protocol for Children Identified as High Risk for Autism in Early Intervention Health Districts
Brief Title: Early Diagnostic Response Model (EDRM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Department of Public Health (Unknown)
Responsible Party: Principal Investigator, Allison Schwartz, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00003763
Record Dates: First submitted 2022-06-09; First posted 2022-06-15 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Autism; Early Intervention; Telehealth; Assessment
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Families with children enrolled in BCW with suspected diagnosis of autism (Experimental): Post-consent, families with children between 16-33 months will receive a link to complete the EAC Developmental History Survey on REDCap and a link to complete parent/caregiver questionnaires about developmental and/or adaptive information. Then, the family will be assigned to a clinician for the autism assessment and scheduled their assessment and feedback session (one week later).
  Interventions: Behavioral: Early Diagnostic Response Model (EDRM)

INTERVENTIONS:
Behavioral: Early Diagnostic Response Model (EDRM) — Use of telehealth capabilities to implement measures and capture and code information related to an autism diagnosis. This program evaluation will be using pre- and post-data and data collected through the process to evaluate the effectiveness of the EDRM pilot.

SUMMARY:
Babies Can't Wait (BCW) in Georgia will be referring families with children seeking an autism spectrum disorder (autism) diagnosis at the Emory Autism Center's (EAC) Child Screening and Assessment Clinic.The objective of this study is to develop, pilot, and evaluate a diagnostic protocol for children identified at high risk for autism in the BCW early intervention program screening (part of a public health service). This program evaluation will be using pre- and post-data and data collected through the process to evaluate the effectiveness of the EDRM pilot.

DETAILED DESCRIPTION:
The objective of this study is to develop, pilot, and evaluate a diagnostic protocol to assess high-risk toddlers for autism spectrum disorder (ASD) diagnosis of families enrolled in the Georgia Babies Can't Wait (BCW) early intervention program. The Early Diagnostic Response Model (EDRM) project will be addressing children who are identified at high risk for ASD according to the BCW screening protocol, which is the M-CHAT-R/F. Community psychologist will be taught the protocol and receive referrals to build capacity and better address the need across the state. Currently, many children who are screening high-risk for ASD in BCW districts are unable to access follow-up evaluations due to limited community resources and long wait times. It is hypothesized that the EDRM will be successful in increasing the number of BCW families that access an ASD evaluation using telehealth tools and testing protocols and that the families and clinicians involved will be satisfied with the streamlined process. The clinicians' conclusions from the EDRM assessment will be based on the Diagnostic and Statistical Manual, 5th edition (DSM-5; American Psychiatric Association [APA], 2013) and are hypothesized to be able to provide high-risk children and their families with the same access to services as an in-person assessment.

A secondary objective is to investigate how many high-risk referral assessments can be completed entirely via streamlined telehealth protocol and how many required additional information to be collected to make a final DSM-5 conclusion.

A tertiary objective is to investigate the improvement of the EDRM as an early identification model to assess for ASD by comparing the numbers of families screened high risk for ASD and referred for an evaluation prior to the study to the number of families who received ASD evaluation by the end of the study through the pilot versus other means. These numbers will be analyzed globally as well as by specific BCW district and other child factors.

ELIGIBILITY:
Inclusion Criteria:

* All families of children between the ages of 16-30 months of age who scored ≥8 on the MCHAT-R and whose BCW provider refers the child to our clinic by 33 months of age will be a possible participant. Evaluations will be done by 36 months of age.
* Referring BCW provider must be one of the participating BCW health districts in this pilot study.
* Parent/Guardian needs to have basic English proficiency
* Parent/Guardian needs to have internet access
* Child must have exposure to English either at home or in out-of-home care (e.g., childcare setting).
* Documentation of M-CHAT-R High-Risk failed score (≥ 8) must be documented in referral.

Exclusion Criteria:

* Families making self-referrals to the EAC or referrals outside of the targeted BCW districts will be excluded from recruitment for this study.
* Children above the age of 33 months at the time of the referral will be excluded as the current EDRM protocol has not been developed in this phase of piloting for individuals over this age.
* Non-English speakers will be excluded from participation due to the current protocol not being applicable to their needs as well as a high correlation between verbal language abilities and social communication and social interaction (SCI) abilities as part of the DSM-5-TR autism criteria.

Ages: 16 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants referred to the Early Diagnostic Response Model (EDRM) | Until the end of the study (approximately one year)
  Monthly numbers of high-risk referrals to the EDRM pilot project and total number of referrals made to the EDRM at the end of the study
Number of participants consented in the Early Diagnostic Response Model (EDRM) study | Monthly until until the end of the study (approximately one year)
  Monthly number of families referred who consent to EDRM participation
Response rate in the Early Diagnostic Response Model (EDRM) study | Until end of the study (approximately one year)
  Response rate will be calculated at project end using the formula [# of families who consented / # of families referred to project] x 100 = response rate)
Number of participants that completed the Early Diagnostic Response Model (EDRM) study | Every 3 months (Quarterly) until end of study (approximately one year)
  Quarterly numbers of participants that completed the EDRM assessment protocol and total number of participants who completed EDRM assessment protocol at study conclusion
Time from referral to completion of the program | Up to 12 weeks post-intervention
  Individual calculation of time from BCW referral to final summary report sent to family using the formula:
  Date of Final Report sent to family - Date of referral from BCW =Time in EDRM pilot

SECONDARY OUTCOMES:
Number of high-risk referral assessments that completed entirely via streamlined telehealth protocol | Every 3 months (Quarterly) until end of study (approximately one year), Up to 12 weeks post-intervention
  Number of high-risk referral assessments that completed entirely via streamlined telehealth protocol, analyzed globally. Monthly, Quarterly, and Total numbers of participants who completed EDRM pilot assessment.
Number of of high-risk referral by BCW district | Every 3 months (Quarterly) until end of study (approximately one year), Up to 12 weeks post-intervention
  Number of high-risk referral assessments by specific BCW district. Monthly, Quarterly, and Total numbers of participants who completed EDRM pilot assessment.
Number of of high-risk referral by child factors | Every 3 months (Quarterly) until end of study (approximately one year), Up to 12 weeks post-intervention
  Number of high-risk referral assessments by child factors. Monthly, Quarterly, and Total numbers of participants who completed EDRM pilot assessment.
Number of of high-risk referral by clinician setting | Every 3 months (Quarterly) until end of study (approximately one year), Up to 12 weeks post-intervention
  Number of high-risk referral assessments by clinician setting. Monthly, Quarterly, and Total numbers of participants who completed EDRM pilot assessment.
Number of participants with additional information collected to make a final DSM-5 conclusion | Every 3 months (Quarterly) until end of study (approximately one year), Up to 12 weeks post-intervention
  Number of participants with additional information collected to make a final DSM-5 conclusion
Parent satisfaction of EDRM assessment survey | At completion of EDRM assessment (4 weeks post-intervention)
  Administered at the end of individual EDRM assessment. Satisfaction surveys will use a Likert-scale of 1-5 with 1 being strongly disagree and 5 being strongly agree as well as 0 being not applicable/unknown. Higher scores indicate more satisfaction with specific aspect of EDRM project.
  Total score: 0 to 110.
BCW provider(s) Service Coordinator satisfaction with EDRM assessment survey | At completion of EDRM assessment (4 weeks post-intervention)
  Administered at end of individual EDRM assessment. Satisfaction surveys will use a Likert-scale of 1-5 with 1 being strongly disagree and 5 being strongly agree as well as 0 being not applicable/unknown. Higher scores indicate more satisfaction with specific aspect of EDRM project.
  Total score: 0 to 110.
Parent satisfaction with access to treatment survey | 3 months after completion of EDRM assessment
  Administered 3-months after completion of EDRM assessment. Satisfaction surveys will use a Likert-scale of 1-5 with 1 being strongly disagree and 5 being strongly agree as well as 0 being not applicable/unknown. Higher scores indicate more satisfaction with specific aspect of EDRM project.
  Total score: 0 to 15.
BCW provider(s) Early Intervention Coordinator satisfaction with EDRM pilot survey | Every 3 months (Quarterly) until end of study (approximately one year), Up to 12 weeks postintervention
  Completed every 3 months (Quarterly). Satisfaction surveys will use a Likert-scale of 1-5 with 1 being strongly disagree and 5 being strongly agree as well as 0 being not applicable/unknown. Higher scores indicate more satisfaction with specific aspect of EDRM project.
  Total score: 0 to 55
Number of families screened high risk for ASD and referred for an evaluation | Through study completion, an average of 1 year
  Number of families screened high risk for ASD and referred for an evaluation
Number of families who received ASD evaluation by the end of the study through the pilot versus other means | Through study completion, an average of 1 year
  Number of families who received ASD evaluation by the end of the study through the pilot versus other means

CONTACTS AND LOCATIONS:
Overall Officials: Allison Schwartz, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the EDRM pilot will be shared, after de-identification process has been completed.
  Proposals may be submitted to up to 3 years following article publication. After 3 years, data will be provided in Emory University's data warehouse but without investigator support other than deposited materials.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of the EDRM pilot project; Beginning 3 months and ending within 3 years of published results through peer-review process.
Access Criteria: Researchers who provide a methodologically sound proposal that has been approved by an IRB. To achieve aims in proposed activity and/or for meta-analysis of telehealth assessments